CLINICAL TRIAL: NCT01569854
Title: An Observational Study Investigating Genetic Influences on Clinical Outcomes and Change in Carotid Intimal Thickness in Adults Taking Atorvastatin, Simvastatin, or Lovastatin
Brief Title: Genetic Influence on Statin Pharmacodynamics
Status: Withdrawn | Type: Observational
Why Stopped: Insufficient recruitment
Sponsor: Ohio State University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Joseph Kitzmiller, Assistant Professor, Ohio State University
Other Study IDs: OSU 2011H0261; K23GM100372 (NIH)
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Hyperlipidemia; Hypercholesterolemia; Dyslipidemia
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — nuclear pellet
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- statin

SUMMARY:
The study intends to investigate whether genetics influence how individuals respond to statins (clinical outcomes and changes in carotid intimal media thickness)

ELIGIBILITY:
Inclusion Criteria:

* recently (within past 3 months) started taking atorvastatin, lovastatin, or simvastatin

Exclusion Criteria:

* concomitant uses of medications, supplements, or OTCs known to interfere with statin metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals will be recruited from various hospitals, ancillary clinics, and primary-care offices affiliated with the Ohio State University Medical Center (OSUMC).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2016-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
carotid intimal media thickness (CIMT) | 2 years
  CIMT measurements will be performed at baseline (within 3 months of starting statin) and at 6, 12, 18, and 24 months. Change in CIMT is considered a surogate measure of atherosclerotic progression.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Kitzmiller, MD PhD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States